CLINICAL TRIAL: NCT03314402
Title: A Randomized, Double-blind,Dose-escalation Phase 1 Study to Assess the Safety, Tolerance, and Pharmacokinetics of Jaktinib,an Oral JAK2 Inhibitor, in Healthy Volunteers
Brief Title: The Tolerance, Pharmacokinetics of Jaktinib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZGJAK001
Record Dates: First submitted 2017-10-10; First posted 2017-10-19 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
Keywords: JAK2 inhibitor; Tolerance; Pharmacokinetics; Dose-escalated

STUDY DESIGN:
Intervention Model Description: SAD: 8 cohorts, 8 subjects take jaktinib and 2 subjects take placebo;
  MAD: 5 cohorts, 8 subjects take jaktinib and 2 subjects take placebo;
  Postprandial Phamocokinetics:12 subjects, crossover designing
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Jaktinib Dihydrochloride Monohydrate
  Interventions: Drug: Jaktinib Dihydrochloride Monohydrate
- group 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Jaktinib Dihydrochloride Monohydrate — Active Substance
  Other Names: Jaktinib
  Arms: group 1
Drug: placebo — Placebo
  Other Names: PLA
  Arms: group 2

SUMMARY:
A randomized, double-blinding, dose-escalated phase 1 trial to evaluate the tolerance and fasting/postprandial pharmacokinetics of jaktinib.

DETAILED DESCRIPTION:
The study is a randomized, double-blind phase 1 trial including 3 independent parts: single ascending dose(SAD) part,multiple ascending dose(MAD) part and postprandial pharmacokinetics part. SAD and MAD are dose-escalated tolerant study designed 8 cohorts and 5 cohorts in SAD and MAD respectively. The aims of the study as below:

1. Evaluating the safety and tolerance of Jaktinib in healthy volunteers.
2. Evaluating the fasting pharmacokinetic parameters of Jaktinib in healthy volunteers.
3. Evaluating the postprandial pharmacokinetic parameters of jaktinib in healthy volunteers.
4. Analysis the metabolites of Jaktinib

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions;
2. Be able to complete the research according to the clinical trial protocol;
3. Subjects (include male subjects) have no pregnancy plan within the next 6 months and voluntarily take effective contraceptive measures;
4. Male and female subjects between 18 and 45 years (inclusive) of age;
5. The weight of a male subject is no lower than 50kg,The female is no lower than 45kg,and having a Body Mass Index (BMI) between 18 to 28 (both inclusive), calculated as weight in kg / height in m2;
6. Health status: no clinical histories with clinical significance about heart, liver, kidney, digestive tract, nervous system, respiratory system (such as asthma), mental disorders and metabolic abnormalities and so on;
7. Physical examination, vital signs normal or no clinical significance.

Exclusion Criteria:

1. Someone smoking more than 5 pieces per day within the 3 months before the trial ；
2. Allergies, such as allergies to Investigational Drug,excipients,or idiosyncratic reaction to drug and food;
3. Having a history of drug and / or alcohol abuse (14 units of alcohol per week: 1 units = beer 285 mL, or 25 mL of spirits, or 100 mL of wine)；
4. Blood donation or extensive blood loss (> 450 mL) within three months of the use of the study drug;
5. Having difficulty of swallowing or any history of gastrointestinal diseases that affect drug absorption;
6. Suffering from any increased risk of hemorrhagic disease, such as hemorrhoids, acute gastritis or gastric and duodenal ulcer, etc.;
7. Taked any drug that changes liver enzyme activity 28 days prior to the use of the study drug;
8. Taked any prescription, OTC drugs, any vitamin products or herbs within 14 days prior to the use of the study drug;
9. Two weeks before the trial took a special diet (including dragon fruit, mango, grapefruit, and / or rich in xanthine diet, etc.) or strenuous exercise, and other activities that affect drug absorption, distribution, metabolism, excretion and so on;
10. Combined with the following CYP3A4, p-gp or Bcrp inhibitors or inducers, such as itraconazole, ketoconazole or dronedarone;
11. There have been significant changes in diet or exercise habits recently;
12. Taked research drugs within three months prior to the use of the study drug or participating in any drug clinical trial;
13. Subjects who were intolerant of high-fat meals (2 boiled eggs, 100g, 20g Bacon, 1 slices of buttered toast, 50g, 115g fries, and 240 ml whole milk) were applied only to subjects who participated in the postprandial test.
14. ECG has clinical significance;
15. Female subjects are in lactation or serum pregnancy test are positive during screening or during the test;
16. Clinical laboratory tests are abnormal and have clinical significance, or other clinical findings showing clinically significant diseases (including but not limited to gastrointestinal, renal, liver, nerves, blood, endocrine, neoplasms, lungs, immunizations, mental or heart Cerebrovascular disease);
17. hepatitis (including hepatitis B and hepatitis C), AIDS, syphilis screening test positive;
18. Acute disease occurs before screening or using test drug;
19. Taking chocolate, any caffeine, or xanthine-rich food or drink at least 48 hours prior to the use of the study drug;
20. Taking any alcoholic products within 24 hours prior to the use of the study drug;
21. Alcohol or drug screening positive or drug abuse history over the past five years or 3 months before the trial used by drug users.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 6 months
  Evaluating Dose-Limiting Toxicities (DLTs) from the individuals taking orally dose-escalated jaktinib

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | up to 120 hours
  The parameter to evaluating the plasma concentration of the oral jaktinib
Area Under the Curve [AUC] | up to 120 hours
  The parameter to evaluating the exposure of the oral jaktinib

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China